CLINICAL TRIAL: NCT03424863
Title: Peak Systolic Blood Pressure in Heart Patients With Aortic Stent-graft During Moderate Intensity Strength Training: A Descriptive Intervention Study
Brief Title: Blood Pressure Changes During Moderate Intensity Strength Training in Aortic Stent-graft Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FYS014
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Aortic Stent Graft

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aortic stent graft patients (Experimental): Patients who have received an aortic stent graft who will perform one session of moderate intensity muscle strengthening during which blood pressure will be measured.
  Interventions: Other: Moderate Intensity Muscle Strengthening
- Healthy volunteers (Experimental): Healthy volunteers in general good health with no history of heart disease who will perform one session of moderate intensity muscle strengthening during which blood pressure will be measured.
  Interventions: Other: Moderate Intensity Muscle Strengthening

INTERVENTIONS:
Other: Moderate Intensity Muscle Strengthening — 1 session of lower extremity muscle strengthening at moderate intensity (60% of estimated maximal muscle strength). The exercise is performed on one single day.

SUMMARY:
Patients with an aortic stent graft are recommended to do muscle strengthening exercise as part of their rehabilitation. But, as excess blood pressure pose a risk to the integrity of the stent graft, high intensity muscle strengthening exercise may potentially be detrimental, and hence moderate intensity muscle strengthening is recommended. However, the blood pressure changes during moderate intensity strengthening exercises are unknown, and this study aims to quantify these among patients and compare them to those of healthy volunteers.

Purpose:

The purpose of this study is to investigate the increase in blood pressure during quadriceps muscle strength training in patients with aortic stent graft.

Methods:

Patients with aortic stent graft will be included. The participants are investigated once. During the investigation, the blood pressure increase during a single strength training exercise (leg press) is measured. The strength training exercise is done at 60% of maximal strength (moderate intensity) corresponding to 15 Repitition Maximum (RM) (a load that can be lifted exactly 15 times).

ELIGIBILITY:
Inclusion Criteria patients:

* Adults (+18y) with aortic stent graft following aortic dissection or aneurism
* Minimum 8 weeks post surgery
* Strengthening exercise approved by treating cardiologist
* Able to perform the exercise

Exclusion Criteria patients:

* Lack of ability to read, speak or understand instructions in Danish or English
* Other unspecified heart disease

Inclusion Criteria healthy volunteers:

* Adults (+18y)
* In good health (self report)

Exclusion Criteria healthy volunteers:

• Lack of ability to read, speak or understand instructions in Danish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Peak systolic pressure during a single lower extremity muscle strengthening exercise | 5 minutes: 15 repetitions of leg press muscle strength exercise.
  Blood pressure is measured continuously using a finger clamp measurement device (Nexfin)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Dall, PhD, Study Chair — Department of Physio- and Occupational Therapy, Bispebjerg-Frederiksberg Hospital, Denmark
Locations (1):
- Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided